CLINICAL TRIAL: NCT04017884
Title: Evaluation of Caries Regression, Color Improvement and Mineral Content of White Spot Lesions Post-orthodontic Treatment After Remineralization With Remin Pro Forte Versus Remin Pro: A Randomized Clinical Trial
Brief Title: Evaluation of Remin Pro Forte Versus Remin Pro on Treatment of White Spot Lesions Post Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mennatallah aboulnaga, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHD-CU-2019-07-10
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: White Spot Lesion
Keywords: Remineralization; caries regression; color improvement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (participant,investigator,outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remin Pro Forte. (Experimental): intervention
  Interventions: Combination Product: Remin Pro
- Remin pro. (Active Comparator): comparator
  Interventions: Combination Product: Remin Pro Forte

INTERVENTIONS:
Combination Product: Remin Pro Forte — a combination of chemicals with natural products cream .
  Arms: Remin pro.
Combination Product: Remin Pro — a combination of chemicals
  Arms: Remin Pro Forte.

SUMMARY:
randomized clinical trial to evaluate caries regression, the change in colour and mineral content of the demineralized enamel after treatment with Remin Pro Forte paste (fluoride, hydroxyapatite, xylitol, ginger, and curcuma) and Remin pro cream which contains (fluoride, hydroxyapatite, xylitol) remineralizing agents with the null hypothesis that Remin Pro forte will have the same clinical performance as Remin Pro in remineralizing white spot lesions post-orthodontic treatment.

DETAILED DESCRIPTION:
Recently, a remineralizing water based cream containing Hydroxyapatite, Fluoride and Xylitol (Remin pro) has been introduced. It has been claimed that hydroxyapatite fills eroded enamel, fluoride seals dentinal tubules and xylitol acts as an antibacterial agents. This product has been assumed to be suitable for management of dentinal hypersensitivity, prevention of enamel demineralization and promoting remineralization of enamel subsurface lesions. There are few studies regarding the effect of calcium phosphate and hydroxyapatite-based agents on remineralization and optical appearance of White spot lesions following orthodontic therapy.

Recently a new formulation of Remin pro has been introduced called (Remin Pro Forte) with the same components of fluoride, hydroxyapatite, xylitol in addition to two natural products (Ginger, curcuma) with the rationale based behind that they have antibacterial effect against streptococcus mutans in addition to anti-cariogenic effect which is being confirmed in the scientific literature.

Follow up period is selected to be 3 months, which is enough for evaluation of the outcomes (caries regression, color change, mineral content) assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. No systemic disease.
2. Has completed fixed orthodontic treatment, brackets debonded.
3. Has at least two teeth with white spot lesion.
4. Has received conventional periodontal therapy after orthodontic treatment.
5. Between the ages of 12 and 25 years of age.

Exclusion Criteria:

1. Presence of enamel hypoplasia or dental fluorosis.
2. Presence of tetracycline pigmentation.
3. Periodontal pocketing of 3mm or greater.
4. Taking antibiotics.
5. Presence of carious cavities.
6. Allergy to fluoride gel / varnish being used in study.
7. Subjects who had evidence of reduced salivary flow or significant tooth wear

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
caries regression | 3 months
  The assessment will be done by photographic image records and performing ICDAS II scoring on white spot lesions on the image records.

SECONDARY OUTCOMES:
color improvement | 3 months
  To assess the color improvement of white spot lesions, Digital photographs of the white spot lesions will be taken using digital camera.

OTHER OUTCOMES:
mineral content | 3 months
  To measure the mineral content of WSLs, the labial surfaces of the selected teeth will be assessed by VistaCam iX using a special head for taking fluorescent images according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: mennatallah aboulnaga, MD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No